CLINICAL TRIAL: NCT06598202
Title: An Exploratory Study on the Use of Intranasal Administration of Small Extracellular Vesicles for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Exploring Nasal Drop Therapy With Small Extracellular Vesicles for ALS
Acronym: de-ALS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Shengqi Medical Technology (Guangzhou) Co., Ltd. (Unknown); Viyun (Xiamen) Biomedical Research Institute Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Junwei Hao, MD, Director of Neurology Department, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XMEC-2024-267-002
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Neurodegenerative diseases; Inflammation; Motor neuron degeneration; Exosomes; Small extracellular vesicles
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exosomes group (Experimental): Patients in this arm will receive exosomes derived from human umbilical cord blood mesenchymal stem cells as a nasal drop, administered once daily, twice a week, for a total of two weeks.
  Interventions: Drug: exosomes derived from human umbilical cord blood mesenchymal stem cells for nasal drop
- Exosomes placebo group (Placebo Comparator): Patients in this arm will receive a placebo nasal drop mimicking exosomes derived from human umbilical cord blood mesenchymal stem cells, administered once daily, twice a week, for a total of two weeks.
  Interventions: Drug: a placebo of exosomes derived from human umbilical cord blood mesenchymal stem cells for nasal drop

INTERVENTIONS:
Drug: exosomes derived from human umbilical cord blood mesenchymal stem cells for nasal drop — Exosomes derived from human umbilical cord blood mesenchymal stem cells for nasal drop (administered once daily, twice a week, for a total of two weeks, based on the recommended dose during the dose-escalation phase).
  Other Names: hUC-MSC-sEV-001
  Arms: Exosomes group
Drug: a placebo of exosomes derived from human umbilical cord blood mesenchymal stem cells for nasal drop — Exosomes placebo
  Other Names: hUC-MSC-sEV-001 placebo
  Arms: Exosomes placebo group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-escalation trial. The goal of this clinical trial is to evaluate the safety and preliminary efficacy of nasal drop exosomes derived from human umbilical cord blood mesenchymal stem cells (hUC-MSC-sEV-001) in amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-escalation trial. The study will consist of two parts: Part 1 will be a dose-escalation study, and Part 2 will be an expanded safety study based on the findings from Part 1.

A traditional 3+3 dose-escalation design will be implemented in Part 1. Cohort 1 will receive low-dose; Cohort 2 will receive middle-dose; and Cohort 3 will receive high-dose. (Cohort 1 to Cohort 3 will receive a dose of 1 mL per nostril, administered once daily, twice a week, for a total of two weeks.) If no dose-limiting toxicities (DLTs) are observed for 2 weeks after the administration of the first nasal drop, a new cohort will be enrolled at the next planned dose level. If DLTs are observed in one participant in the cohort, an additional three participants will be treated at the same dose level. Dose escalation will be stopped if DLTs are observed in more than 33% of the participants.

In Part 2, 20 subjects will be randomized in a 1:1 ratio [exosome (n=10) or exosome placebo (n=10)]. The dose level will be determined by the primary researcher based on the findings from Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years, inclusion of both genders;
* Disease duration: ≥6 months and ≤2 years (counted from the onset of any ALS symptoms);
* Subjects must meet the El Escorial revised criteria (2000) for the diagnosis of ALS, with a diagnosis of Definite ALS, Probable ALS, Probable laboratory-supported ALS, or Possible ALS;
* A score of ≥2 on each item of the revised ALS Functional Rating Scale (ALSFRS-R), with a score of 4 for items related to dyspnea, orthopnea, and respiratory insufficiency;
* BMI: Between 18 and 30 kg/m²;
* Subjects must have a baseline forced vital capacity percentage (%FVC) ≥70%;
* Allowed concomitant treatments: Oral administration of riluzole/edaravone at standard doses for ≥30 days; regular intravenous edaravone with planned sequential oral treatment. During the trial and follow-up period, the dosage and type of concomitant medications must remain unchanged;
* Subjects of childbearing potential must use appropriate and effective contraception from 2 weeks prior to trial enrollment until the end of the follow-up period;
* The subject or legal representative must be able to sign an informed consent form and comply with the study requirements for medication administration and follow-up.

Exclusion Criteria:

* Diagnosed as non-ALS based on clinical presentation and available clinical examinations (e.g., neurophysiological tests, MRI, or other imaging, laboratory tests);
* Abnormal nasal anatomy, nasal cavity damage, severe rhinitis, or nasal disease affecting the administration of the study drug;
* Requires nasal insertion of a gastric tube;
* Peripheral venous hemoglobin (HGB) < 100 g/L, absolute neutrophil count (NEUT) < 1.5×10^9/L, platelet count (PLT) < 100×10^9/L, white blood cell count (WBC) < 4.0×10^9/L or ≥ 12×10^9/L, serum albumin < 30 g/L; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3× the upper limit of normal (ULN);
* Severe renal insufficiency: Glomerular Filtration Rate (GFR) < 30 mL/min (Cockcroft-Gault formula), or other known severe renal diseases;
* Positive for hepatitis B surface antigen, e antigen, e antibody, or core antibody combined with positive hepatitis B virus DNA; positive for hepatitis C virus antibody; positive syphilis serum antibody; or positive for HIV antibody;
* History of acute myocardial infarction or interventional treatment within the last 6 months, or heart failure (classified as NYHA III-IV);
* Presence of severe localized or systemic infection, immunodeficiency, or currently taking immunosuppressants;
* Concurrent severe systemic diseases such as immunodeficiency diseases, coagulation disorders, or malignancies;
* Vaccination within 1 month prior to the first administration or during the study until the end of follow-up;
* Known allergy to the drugs used in this study or similar drugs;
* Participation in another study and administration of an investigational product within the last 3 months;
* Contraindications to MRI (e.g., presence of metal implants) or inability to tolerate MRI (e.g., claustrophobia);
* Pregnant or breastfeeding women, or women of childbearing potential who cannot or are unwilling to use appropriate contraception;
* Unwillingness or inability to comply with the procedures required by the protocol;
* Any other conditions deemed unsuitable for inclusion by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced dose-limiting Toxicities (DLTs) | 24 hours, 4±1 Weeks
  DLTs related to hUC-MSC-sEV-001 include adverse events of grade 3 or higher (including significant clinical laboratory findings) that are possibly, likely, or definitely related to the study drug, accompanied by clinical symptoms and requiring medical treatment within 14 days of administration. Adverse events are graded according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0).

SECONDARY OUTCOMES:
Incidence of severe adverse events | 4±1 Weeks
  The proportion of patients who experienced severe adverse events.
Change from baseline in ALS functional rating scale - revised | 4±1 Weeks, 12±1 Weeks, 24±1 Weeks
  The ALSFRS-R is rating scale (ratings 0 = can't do, to 4 = normal ability) used to determine participants' assessment of their capability and independence in 12 functional activities.
  This is a validated scale, both in person and by phone, which provides a total score from four sub-scores which assess speech and swallowing (bulbar function), use of upper extremities (cervical function), gait and turning in bed (lumbar function), and breathing (respiratory function).
  Total scores range from 0 (most impaired) to 48 (normal ability).
Change from baseline in forced vital capacity to predicted value ratio (FVC% pred) | 4±1 Weeks, 24±1 Weeks
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced vital capacity (FVC) is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration.
Time to event (death, tracheostomy, and permanent assisted mechanical ventilation) | up to 24 Weeks
  The number of time-to-event outcomes.
Change from baseline in the Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40). | 4±1 Weeks, 12±1 Weeks, 24±1 Weeks
  ALSAQ-40 score ranges from 0 to 160 points, and higher scores indicate better quality of life.
Change from baseline in the Edinburgh Cognitive and Behavioral ALS Screen (ECAS). | 12±1 Weeks, 24±1 Weeks
  ECAS determine cognitive and behavioral changes of patients suffering from Amyotrophic Lateral Sclerosis.
  With ECAS, ALS-specific (fluency, executive functions and social cognition, language; minimum score = 0, maximum score = 100) and ALS-nonspecific (memory, visuospatial functions; minimum score = 0, maximum score = 36) functions can be analyzed to enable the distinction from other diseases with cognitive and behavioral impairments.
Change from baseline in the Neurophysiological Index (NI) and Compound Muscle Action Potential (CMAP) score. | 12±1 weeks
  The NI is derived from the CMAP, the DML and the F-wave frequency (CMAP amplitude/DML) x F frequency %), representing aspects of the effects of denervation and reinnervation, of degeneration of the terminal part of the motor axons, and of the excitability of anterior horn cells.
  The negative amplitudes of the CMAP for motor nerve conduction in the median and ulnar nerves in the upper extremities as well as the peroneal and tibial nerves in the lower extremities of ALS patients were recorded (median nerve-wrist, ulnar-wrist, peroneal-ankle, tibial-ankle). These nerves were scored based on the decrease in the amplitudes of each nerve CMAP- 0 (CMAP> =[X-2s]), 1 (50% [X-2s] < CMAP < [X-2s]), 2 (30% [X-2s] < CMAP < 50% [X-2s]), 3 (CMAP < =30% [X-2s]), respectively. The values of X and S for different nerves and different patient age groups, which were applied in the electrophysiology examination room.
Change from baseline in the Rasch Overall ALS Disability Scale (ROADS). | 4±1 Weeks, 12±1 Weeks, 24±1 Weeks
  ROADS score ranges from 0 to 56 points, and higher scores indicate better basic daily function.
Change from baseline in the Medical Research Council (MRC) Scale. | 4±1 Weeks, 12±1 Weeks, 24±1 Weeks
  MRC ranges from 0 to V grades, and higher grades indicate higher muscle strength.
Change from baseline in the the Lower Motor Neuro Scale(LMNS). | 4±1 Weeks, 12±1 Weeks, 24±1 Weeks
  LMNS was calculated using the score proposed by Devine et al. that assign a separate LMN score for each limb, ranging from 0 (no involvement) to 3 (significant, severe involvement), based on the Medical Research Council and muscle wasting.

OTHER OUTCOMES:
Change from baseline in the neuroimaging indices. | 24±1 weeks
  Neuroimaging indices include gray matter thickness, gray matter volume, white matter volume, DTI metrics of the corticospinal tract, DTI-ALPS, and QSM of the bilateral motor cortex.
Change from baseline in the blood markers. | up to 24 weeks
  A number of blood markers will be examined including C-reactive protein, neurofilament light chain, IL-1β, IL-6, IL-8, IL-10, Tumor Necrosis Factor-alpha.

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD; PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital ,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data to other researchers.